CLINICAL TRIAL: NCT05087043
Title: Effects of Oral Stimulation and Supplemental Nursing System on the Transition Time to Full Breast of Mother and Sucking Success in Preterm Infants
Brief Title: Effects of Oral Stimulation and Supplemental Nursing System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Gonca Karayagiz Muslu, Faculty of Fethiye Health Science, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1
Record Dates: First submitted 2021-09-15; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Breastfeeding
Keywords: Preterm; oral stimulation; supplemental nursing system
MeSH Terms: conditions — Breast Feeding; Premature Birth

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Stimulation and Supplemental Nursing System group (Experimental): Oral motor Stimulation (OMS) and an Supplemental Nursing System (SNS) were applied to preterm infants in the experimental group.
  Interventions: Device: Oral motor stimulation (OMS) and The supplemental nursing system (SNS)
- control group (No Intervention): The clinic's routine feeding protocol was applied to the babies in the control group.

INTERVENTIONS:
Device: Oral motor stimulation (OMS) and The supplemental nursing system (SNS) — OMS and an SNS were applied to preterm infants in the experimental group. Oral stimulation intervention provides assisted movement to activate muscle contraction and provides movement against resistance to build strength. The cheeks (internal and external), lips, gums, tongue, and palate were stimulated by finger-stroking following the protocol. OMS consisted of intra (oral region) and peri-oral stimulation (around the oral region). The OMS was administered three times a day by a nurse, from the day of initiation of oral feeding to the day of independent oral feeding 15 minutes before the feeding schedule. A bottle/container was filled with breast milk before the process and given to the baby via SNS while the baby was holding the mother's breast. The SNS consists of a syringe/container and a feeding catheter. One end of the feeding probe is inside the syringe/container, while the other end of it is fixed to the mother's nipple using plaster.
  Arms: Oral Stimulation and Supplemental Nursing System group

SUMMARY:
This study aimed to investigate the effect of oral stimulation and a supplemental nursing system on the time to full maternal breastfeeding and sucking success in preterm infants.

DETAILED DESCRIPTION:
This study aimed to investigate the effect of oral stimulation and a supplemental nursing system on the time to full maternal breastfeeding and sucking success in preterm infants. The sample consisted of 70 preterm babies. Oral motor stimulation and a supplemental nursing system were applied to the preterm infants in the experimental group, while no intervention was applied to those in the control group.

ELIGIBILITY:
Inclusion Criteria:

* a birth weight of 1,000 gr and above,
* a gestational age between 30 and 34 weeks,
* no congenital anomaly,
* no severe asphyxia or chronic lung disease,
* spontaneous breathing,
* grades III and IV intracranial hemorrhage and no periventricular leukomalacia

exclusion criteria.

* congenital anomaly
* grades III and IV intracranial hemorrhage and periventricular leukomalacia

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
transition times to oral feeding | up to three weeks
  Transition time to oral feeding is the time that the preterm baby outgrew gavage feeding and fed with complementary nutritional support, and it was evaluated as days in the study.
transition times to full breast | up to 15 days
  The transition time to full breastfeeding is the duration from the day that the preterm baby started oral nutrition until the day they started breastfeeding
the weight of the babies when they started oral nutrition | up to three weeks
  . The oral nutrition body weight is the weight of preterm babies when they started oral nutrition after gavage.
the weight of the babies when they started full breastfeeding | up to 15 days
  The full breastfeeding body weight is the weight in grams of preterm babies when they started feeding from the breast alone
the duration of the baby's discharge | up to 2 months
  The duration of discharge is the number of days between the admission of preterm babies to intensive care and their discharge
The oral nutrition body weight | up to three weeks
  The oral nutrition body weight is the weight of preterm babies when they started oral nutrition after gavage.
The full breastfeeding body weight | up to 15 days
  The full breastfeeding body weight is the weight in grams of preterm babies when they started feeding from the breast alone.
The discharge body weight | up to 2 months
  The discharge body weight is the weight in grams of preterm babies at discharge
The sucking success | In the first month after discharge
  The sucking score of preterm babies was determined using LATCH breastfeeding scores at discharge.

SECONDARY OUTCOMES:
Heart rate of the babies | 15 minutes
  Heart rate
respiratory rate of the babies | 15 minutes
  respiratory rate
oxygen saturation of the babies | 15 minutes
  oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: gonca muslu, Study Chair — Muğla Sıtkı Koçman University
Locations (1):
- Gonca Muslu, Fethiye, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT05087043/Prot_SAP_000.pdf